CLINICAL TRIAL: NCT05162378
Title: Impact of Treatment With Amotosalen on the Practice of Platelet Transfusion in Adult Heart Surgery
Brief Title: Amotosalen and Platelet Transfusion in Adult Heart Surgery
Acronym: TransAdult
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7994
Record Dates: First submitted 2021-10-12; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-10

CONDITIONS: Heart Surgery
Keywords: Amotosalen; Platelet transfusion; Bleeding; heart surgery
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Blood safety is ensured by the rigorous selection of donors and biological tests. However, infectious agents can escape this detection and be transmitted to recipients during transfusion. Amotosalen is a derivative of psoralens that intercalates with nucleic acids and inactivates them after UV exposure; it therefore makes it possible to inhibit any replication of an infectious agent present. Preliminary studies have shown its safety and efficacy in preventing the transmission of infectious agents during the administration of labile blood products (fresh frozen plasma and platelet concentrates) as well as the absence of loss of efficacy (absence of loss of pro-aggregating and procoagulant properties) of the transfused products. In addition, there is a significant reduction in side effects for platelet concentrates, especially compared to irradiated concentrates.

Treatment of platelet concentrates with Amotosalen may be responsible for a reduction in the platelet concentration in each concentrate with an overall decrease in efficiency and transfusion yield compared to untreated concentrates.

ELIGIBILITY:
Inclusion criteria:

* Major subjects ≥18 years old
* Cardiac surgery or ascending aorta
* Platelet transfusion for any reason
* Subject not having expressed their opposition, after information, to the reuse of their data for the purposes of this research

Exclusion criteria

* Subject having expressed opposition to participating in the study
* Presence or - installation of transient circulatory assistance (outside of the CEC) or definitive
* Heart or cardiopulmonary transplantation
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subjects having had cardiac surgery or ascending aorta and platelet transfusion for any reason
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of the impact of the treatment with Amotosalen on the platelet transfusion practice in adult cardiac surgery unit | Files analysed retrospectively from January 01, 2016 to June 30, 2019 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DELABRANCHE, MD, Principal Investigator — Service d'Anesthésie et Réanimation chirurgicale - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service d'Anesthésie et Réanimation chirurgicale - Hôpitaux Universitaires de Strasbourg, Strasbourg, France